CLINICAL TRIAL: NCT03697499
Title: Effects of Fish Oil in Alleviating Cardiopulmonary Hazards Associated With Ozone Exposure in Young Healthy Adults
Brief Title: Effects of Fish Oil in Alleviating Health Hazards Associated With Ozone Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, PhD and Professor, Fudan University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: FDUEH-4
Record Dates: First submitted 2018-09-30; First posted 2018-10-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular System; Respiratory System; Oxidative Stress; Inflammation
Keywords: ozone exposure; fish oil; 2*2 factorial design
MeSH Terms: conditions — Inflammation | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fish oil and acute ozone exposure (Experimental): The participants will take fish oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour ozone exposure (200 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Interventions: Combination Product: fish oil and acute ozone exposure
- fish oil and shame exposure (Sham Comparator): The participants will take fish oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour shame exposure (0 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Interventions: Combination Product: fish oil and sham exposure
- soy oil and acute ozone exposure (Placebo Comparator): The participants will take soy oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour ozone exposure (200 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Interventions: Combination Product: soy oil and acute ozone exposure
- soy oil and shame exposure (Other): The participants will take soy oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour shame exposure (0 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Interventions: Combination Product: soy oil and sham exposure

INTERVENTIONS:
Combination Product: fish oil and acute ozone exposure — The participants will take fish oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour ozone exposure (200 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Arms: fish oil and acute ozone exposure
Combination Product: fish oil and sham exposure — The participants will take fish oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour shame exposure (0 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Arms: fish oil and shame exposure
Combination Product: soy oil and acute ozone exposure — The participants will take soy oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour ozone exposure (200 ppb ozone) will be conducted in a chamber after four weeks of supplementation.
  Arms: soy oil and acute ozone exposure
Combination Product: soy oil and sham exposure — The participants will take soy oil (2.2 g/day, two 1.1-g capsules daily) in divided doses. Two hour shame exposure (0 ppb ozone) will be conducted in a chamber after four weeks of supplementation
  Arms: soy oil and shame exposure

SUMMARY:
This study aims to evaluate whether dietary supplementation with fish oil can protect against the cardiopulmonary effects induced by ozone exposure.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial among 64 healthy young adults in Shanghai, China. The eligible participants will be randomly assigned in a 2*2 factorial design to 1 of 4 groups: 1) fish oil and ozone exposure, 2) fish oil and shame exposure, 3) soy oil and ozone exposure, or 4) soy oil and shame exposure. The participants who take fish oil would receive 2.2 g/day (two 1.1-g capsules daily) in divided doses, and other participants will take the same amount of soy oil capsules. Two hour ozone exposure (200 ppb ozone) or shame exposure (0 ppb ozone) will be conducted in a chamber after four weeks of supplementation. Ozone is generated by a silent electric discharge method (HTU-500, AZCO Industries Ltd., Canada) and introduced into the chamber. The temperature and relative humidity in the chamber are maintained at 22±1℃ and 50%±5%, respectively. During the 2-hour exposure, each subject alternate 15 minutes of exercise on a treadmill and 15 minutes of rest. The exercise workload would be adjusted to achieve the targeted ventilation of 20±1 L/min/m2 body surface area. Health examinations will be conducted immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during study period;
* Ability to complete the training exercise to induce an inspired ventilation rate of 20±1 L/min/m2 body surface area;
* Body mass index >18.5 and ≤30 (30 is the lower limit for class 2 obesity for Chinese);
* Taking the fish oil or placebo on time.

Exclusion Criteria:

* Being allergic to seafood;
* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic disease, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular disease, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory disease, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic disease, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects with a history of major surgery;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Abnormal baseline 12-lead resting electrocardiogram;
* Abnormal blood index, such as cell counting, blood lipids, and glutamic-pyruvic transaminase (GPT).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Changes of FEV1 | FEV1 will be examined immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning
  Changes of forced expiratory volume in 1 second
Changes of FVC | FVC will be examined immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning
  Changes of forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Principal Investigator — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided